CLINICAL TRIAL: NCT00560560
Title: A Phase II, Single Arm Study Of CP-751,871 In Patients With Refractory Metastatic Adenocarcinoma Of The Colon Or Rectum
Brief Title: Study Using CP-751,871 In Patients With Stage IV Colorectal Cancer That Has Not Responded To Previous Anti-Cancer Treatments
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A4021006
Record Dates: First submitted 2007-11-15; First posted 2007-11-19 (Estimated); Results first posted 2013-05-09 (Estimated); Last update posted 2013-05-20 (Estimated); Status verified 2013-05

CONDITIONS: Colorectal Neoplasm
Keywords: Refractory Colorectal; Single arm; Phase 2
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): Single arm study
  Interventions: Biological: CP-751, 871

INTERVENTIONS:
Biological: CP-751, 871 — Human IgG2 Monoclonal Antibody. 20mg/kg or 30 mg/kg every 3 weeks for 17 cycles, until progression or unacceptable toxicity develops.

SUMMARY:
This study will test if there is any survival benefit in patients with refractory metastatic colorectal cancer that receive CP-751, 871.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have stage IV colorectal cancer
* Patients whose disease has worsened despite prior anti-cancer therapy
* Patients who have satisfactory bonemarrow, kidney and liver function

Exclusion Criteria:

* Patients who are being simultaneously treated with another anti-cancer therapy.
* Patients who have previously received anti-cancer therapy that works like CP-751, 871 (targets insulin-like growth factor receptor)
* Patients that are pregnant or breast-feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 168 (Actual)
Dates: Start 2007-12; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (12):
- United States (2):
  - Pfizer Investigational Site, San Francisco, California
  - Pfizer Investigational Site, Dallas, Texas
- Spain (4):
  - Pfizer Investigational Site, Elche, Alicante
  - Pfizer Investigational Site, Barcelona, Barcelona
  - Pfizer Investigational Site, L'Hospitalet de Llobregat, Barcelona
  - Pfizer Investigational Site, Seville, Sevilla
- United Kingdom (6):
  - Pfizer Investigational Site, Peterborough, Cambridgeshire
  - Pfizer Investigational Site, Leicester, Leicestershire
  - Pfizer Investigational Site, Cardiff
  - Pfizer Investigational Site, Glasgow
  - Pfizer Investigational Site, Peterborough
  - Pfizer Investigational Site, Southampton

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A4021006&StudyName=Study%20Using%20CP-751%2C871%20In%20Patients%20With%20Stage%20IV%20Colorectal%20Cancer%20That%20Has%20Not%20Responded%20To%20Previous%20Anti-Cancer%20Treatments

RESULTS

PARTICIPANT FLOW:
Groups:
- Figitumumab 20 mg/kg: Figitumumab (CP-751,871) was given in 3-week cycles for a total of up to 17 cycles. Participants can receive treatment beyond 17 cycles provided clinical benefit is being achieved. Figitumumab 20 milligram/kilogram (mg/kg) was administered as an intravenous (IV) infusion on Day 1 and 2 in Cycle 1 (loading dose), and on Day 1 of every cycle thereafter.
- Figitumumab 30 mg/kg: Figitumumab (CP-751,871) was given in 3-week cycles for a total of up to 17 cycles. Participants can receive treatment beyond 17 cycles provided clinical benefit is being achieved. Figitumumab 30 milligram/kilogram (mg/kg) was administered as an IV infusion on Day 1 and 2 in Cycle 1 (loading dose), and on Day 1 of every cycle thereafter.
Period: Overall Study
Arm/Group | Figitumumab 20 mg/kg | Figitumumab 30 mg/kg
Started | 85 | 83
Completed | 0 | 0
Not Completed | 85 | 83

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Figitumumab 20 mg/kg | Figitumumab 30 mg/kg | Total
Number analyzed (Participants) | 85 | 83 | 168
Age, Customized [Number; unit: participants]
  <65 years | 56 | 59 | 115
  >=65 years | 29 | 24 | 53
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 39 | 35 | 74
  Male | 46 | 48 | 94

OUTCOME MEASURES:

1. Primary Outcome: Estimate of the 6 Month Survival Probability
Description: The 6 month survival probability was defined as the probability of survival at 6 months based on the Kaplan-Meier estimate. The time was from date of enrollment to date of death due to any cause. For participants who were last known to be alive, overall survival was censored at the last contact date.
Time Frame: Baseline up to Month 6
Population: All enrolled participants.
Measure: Number (95% Confidence Interval); unit: Percent chance of survival
Arm/Group | Figitumumab 20 mg/kg | Figitumumab 30 mg/kg
Number analyzed (Participants) | 85 | 83
Percent chance of survival | 49.4 [38.8 to 60.0] | 44.1 [33.4 to 54.9]
Statistical Analysis 1: Comparison: Figitumumab 20 mg/kg vs Figitumumab 30 mg/kg; The hypotheses for each group were H0:p=0.45 vs H1:p>0.45. There was one interim analysis for futility for each group based on the method of Case and Morgan. The futility boundary was not crossed for 20/kg mg group, but was crossed for the 30/kg mg group. It was recommended to investigators that participants be discontinued from treatment with 30 mg/kg of figitumumab; Test type: Superiority or Other; p > 0.05, Test of probability of 6 month survival — The final analysis was intended to be a binomial test (death prior to 6 months, yes or no). However, 2 participants in the 30/kg mg group were censored prior to 6 months, so the six month Kaplan and Meier estimates were used for each group instead; p-Value >0.05 applies to each group (20 mg/kg and 30 mg/kg). Greenwood's formula was used for standard deviation

2. Secondary Outcome: Overall Survival
Description: The time from date of enrollment to date of death due to any cause. For participants who were last known to be alive, overall survival was censored at the last contact date.
Time Frame: From date of enrollment until death or censorship, up to 33 months
Population: All enrolled participants.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Figitumumab 20 mg/kg | Figitumumab 30 mg/kg
Number analyzed (Participants) | 85 | 83
Months | 5.8 [4.3 to 7.1] | 5.6 [4.1 to 6.9]

3. Secondary Outcome: Progression-Free Survival (PFS)
Description: The period from study entry until disease progression. Participants without progression or death were censored at time of last disease assessment. Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0), as 20% increase in the sum of longest diameters of target measurable lesions, or a clear increase in a non-target lesion, or the apprearance of new lesions.
Time Frame: Baseline until tumor progression or censorship, up to 33 months. The frequency of tumor assessments was screening, every cycle, end of treatment (within 28 days of last dose of study drug), and follow-up.
Population: All enrolled participants.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Figitumumab 20 mg/kg | Figitumumab 30 mg/kg
Number analyzed (Participants) | 85 | 83
months | 1.4 [1.3 to 1.8] | 1.4 [1.3 to 1.7]

4. Secondary Outcome: Percentage of Participants With Objective Response
Description: Percentage of participants with OR based assessment of confirmed complete response (CR) or confirmed partial response (PR) according to Response Evaluation Criteria in Solid Tumors (RECIST). CR was defined as complete disappearance of all target and non-target disease. PR applied only to participants with at least one measurable lesion. Greater than or equal to 30 % decrease under baseline of the sum of longest diameters of all target measurable lesions.
Time Frame: Baseline, every cycle (Day 15-21 or according to local standard), end of treatment (within 28 days of last dose of study drug) and follow-up (150 days after last dose of study drug), up to 33 months
Population: Per protocol. All enrolled participants who started treatment, with measurable disease and adequate baseline assessment.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Figitumumab 20 mg/kg | Figitumumab 30 mg/kg
Number analyzed (Participants) | 75 | 81
Percentage of participants | 0 [0.0 to 4.8] | 0 [0.0 to 4.5]

5. Secondary Outcome: Descriptive Summary of Figitumumab Concentration Versus Time
Description: The measurement of mean plasma concentration of figitumumab in Day 1 of Cycle 1,2,3,4,5
Time Frame: Pre-dose on Day 1, 1 hour after end of infusion (post-dose) on Day 2 in Cycle 1, pre-dose on Day 1 in Cycles 2,3,4, 1 hour post-dose on Day 1 in Cycle 5
Population: All participants for whom PK was assessed at least once. The numbers of participants analyzed are numbers of observation (non-missing concentrations). The numbers for 20 mg/kg group are 84,7,3,2,13 for five cycles, respectively. The numbers for 30 mg/kg group are 79,8,2,2,8 for five cycles, respectively.
Measure: Mean (Standard Deviation); unit: miligrams/liter (mg/L)
Arm/Group | Figitumumab 20 mg/kg | Figitumumab 30 mg/kg
Number analyzed (Participants) | 85 | 83
miligrams/liter (mg/L)
  Cycle1/Day2 | 647.0 (288.23) | 877.7 (230.22)
  Cycle2/Day1 | 244.0 (114.00) | 221.0 (119.65)
  Cycle3/Day1 | 255.7 (60.476) | 245.0 (19.799)
  Cycle4/Day1 | 76.30 (1.2728) | 427.0 (86.267)
  CYcle5/Day1 | 756.2 (239.08) | 745.5 (216.14)

6. Secondary Outcome: Participants Reporting Positive for Total Anti-drug Antibodies (ADA)
Description: The immunogenicity of figitumumab in terms of producing an antidrug antibody (ADA) response were monitored.
Time Frame: Up to 2 hours prior to infusion in Cycles 1 and 4, at the end of treatment, and at the 4th scheduled follow-up visit (~150 days after the last infusion)
Population: Participants for whom at least one ADA measurement was done. The outcome was not analyzed and only listing of ADA level for each participant was available.
Arm/Group | Figitumumab 20 mg/kg | Figitumumab 30 mg/kg
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Counts of Circulating Tumor Cells (CTCs) Expressing Positive Insulin-like Growth Factor 1 Receptor (IGF-1R)
Description: The quantification of circulating tumor cells (CTCs) expressing the IGF-1R in this patient population. Blood samples were collected, and were measured using an automated microscope system.
Time Frame: Cycle 1 pre-dosing and Cycle 4 pre-dosing
Population: All enrolled participants who started treatment and who have at least one sample submitted. The total number of participants for this outcome measure was less than the original population. "N" means the numbers of units analyzed in Pre-treatment and/or Baseline, and Post-Baseline and/or Follow-up, respectively.
Measure: Median (Standard Deviation); unit: number of CTC expressing IGF-1R/ml blood
Arm/Group | Figitumumab 20 mg/kg | Figitumumab 30 mg/kg
Number analyzed (Participants) | 85 | 83
number of CTC expressing IGF-1R/ml blood
  Pre-treatment and/or baseline (n=44,71) | 2.02 (8.79) | 0.54 (1.29)
  Post-Baseline and/or follow-up (n=18,17) | 0.22 (0.55) | 0.00 (0.00)

8. Secondary Outcome: Counts of Circulating Tumor Cells (CTCs)
Description: The quantification of circulating tumor cells (CTCs)in this patient population. Blood samples were collected, and were measured using an automated microscope system.
Time Frame: Cycle 1 pre-dosing and Cycle 4 pre-dosing
Population: as for outcome 7
Measure: Median (Standard Deviation); unit: Number of CTC/ml of blood
Arm/Group | Figitumumab 20 mg/kg | Figitumumab 30 mg/kg
Number analyzed (Participants) | 85 | 83
Number of CTC/ml of blood
  Pre-treatment and/or baseline (n=44,71) | 7.25 (16.59) | 4.90 (9.83)
  Post-Baseline and/or follow-up (n=19,17) | 1.26 (1.94) | 2.18 (7.06)

ADVERSE EVENTS:
Time Frame: Includes date up to 150 days after last dose of study drug
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | Figitumumab 20 mg/kg | Figitumumab 30 mg/kg
Serious Adverse Events (participants affected / at risk) | 56/85 | 53/83
Other Adverse Events (participants affected / at risk) | 85/85 | 83/83
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Figitumumab 20 mg/kg (N=85) | Figitumumab 30 mg/kg (N=83)
Anaemia (Blood and lymphatic system disorders) | 3 | 1
Neutropenia (Blood and lymphatic system disorders) | 2 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 2
Constipation (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 4 | 4
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 2 | 2
Proctalgia (Gastrointestinal disorders) | 1 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 1
Vomiting (Gastrointestinal disorders) | 2 | 4
Coagulopathy (Blood and lymphatic system disorders) | 0 | 1
Heparin-induced thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1
Deafness bilateral (Ear and labyrinth disorders) | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1
Ascites (Gastrointestinal disorders) | 0 | 1
Gastrointestinal perforation (Gastrointestinal disorders) | 0 | 1
Disease progression (General disorders) | 49 | 43
Fatigue (General disorders) | 1 | 0
General physical health deterioration (General disorders) | 2 | 3
Malaise (General disorders) | 1 | 0
Oedema peripheral (General disorders) | 1 | 0
Ulcer (General disorders) | 1 | 0
Asthenia (General disorders) | 0 | 2
Pyrexia (General disorders) | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 0 | 1
Hepatic pain (Hepatobiliary disorders) | 0 | 1
Infection (Infections and infestations) | 1 | 2
Klebsiella bacteraemia (Infections and infestations) | 1 | 0
Lower respiratory tract infection (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 1 | 1
Pyelonephritis (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 3 | 1
Abdominal sepsis (Infections and infestations) | 0 | 1
Bacteraemia (Infections and infestations) | 0 | 1
Escherichia infection (Infections and infestations) | 0 | 1
Spinal cord injury cauda equina (Injury, poisoning and procedural complications) | 1 | 0
Fracture (Injury, poisoning and procedural complications) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 3
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 0
Cerebral haemorrhage (Nervous system disorders) | 1 | 0
Cognitive disorder (Nervous system disorders) | 1 | 0
Dizziness (Nervous system disorders) | 1 | 0
Lethargy (Nervous system disorders) | 2 | 0
Headache (Nervous system disorders) | 0 | 1
Transient ischaemic attack (Nervous system disorders) | 0 | 1
Confusional state (Psychiatric disorders) | 1 | 3
Renal failure (Renal and urinary disorders) | 1 | 0
Renal failure acute (Renal and urinary disorders) | 3 | 2
Hydronephrosis (Renal and urinary disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Figitumumab 20 mg/kg (N=85) | Figitumumab 30 mg/kg (N=83)
Anaemia (Blood and lymphatic system disorders) | 9 | 6
Neutropenia (Blood and lymphatic system disorders) | 4 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 3
Coagulopathy (Blood and lymphatic system disorders) | 0 | 1
Heparin-induced thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1
Palpitations (Cardiac disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 1
Tachycardia (Cardiac disorders) | 0 | 1
Cerumen impaction (Ear and labyrinth disorders) | 1 | 0
Deafness (Ear and labyrinth disorders) | 2 | 2
Hypoacusis (Ear and labyrinth disorders) | 2 | 2
Tinnitus (Ear and labyrinth disorders) | 1 | 0
Vertigo (Ear and labyrinth disorders) | 1 | 0
Deafness bilateral (Ear and labyrinth disorders) | 0 | 1
Deafness unilateral (Ear and labyrinth disorders) | 0 | 1
Ear pain (Ear and labyrinth disorders) | 0 | 1
Motion sickness (Ear and labyrinth disorders) | 0 | 1
Abdominal distension (Gastrointestinal disorders) | 1 | 1
Abdominal pain (Gastrointestinal disorders) | 14 | 11
Abdominal pain lower (Gastrointestinal disorders) | 4 | 2
Abdominal pain upper (Gastrointestinal disorders) | 8 | 7
Anal inflammation (Gastrointestinal disorders) | 1 | 0
Cheilitis (Gastrointestinal disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 17 | 0
Diarrhoea (Gastrointestinal disorders) | 15 | 25
Dry mouth (Gastrointestinal disorders) | 2 | 1
Dyspepsia (Gastrointestinal disorders) | 2 | 6
Dysphagia (Gastrointestinal disorders) | 1 | 1
Faeces discoloured (Gastrointestinal disorders) | 1 | 0
Flatulence (Gastrointestinal disorders) | 2 | 1
Gastrointestinal disorder (Gastrointestinal disorders) | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Gingivitis (Gastrointestinal disorders) | 1 | 0
Glossodynia (Gastrointestinal disorders) | 1 | 0
Intestinal obstruction (Gastrointestinal disorders) | 3 | 1
Mucous stools (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 23 | 27
Oesophagitis (Gastrointestinal disorders) | 1 | 0
Proctalgia (Gastrointestinal disorders) | 1 | 3
Rectal haemorrhage (Gastrointestinal disorders) | 2 | 3
Rectal tenesmus (Gastrointestinal disorders) | 1 | 1
Salivary hypersecretion (Gastrointestinal disorders) | 1 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 1
Stomatitis (Gastrointestinal disorders) | 1 | 3
Tongue disorder (Gastrointestinal disorders) | 1 | 1
Toothache (Gastrointestinal disorders) | 1 | 2
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 1
Vomiting (Gastrointestinal disorders) | 21 | 16
Abdominal discomfort (Gastrointestinal disorders) | 0 | 1
Ascites (Gastrointestinal disorders) | 0 | 1
Gastric atony (Gastrointestinal disorders) | 0 | 1
Gastritis (Gastrointestinal disorders) | 0 | 1
Gastrointestinal perforation (Gastrointestinal disorders) | 0 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 2
Gingival bleeding (Gastrointestinal disorders) | 0 | 1
Gingival disorder (Gastrointestinal disorders) | 0 | 1
Haematochezia (Gastrointestinal disorders) | 0 | 1
Melaena (Gastrointestinal disorders) | 0 | 1
Mouth haemorrhage (Gastrointestinal disorders) | 0 | 1
Oral pain (Gastrointestinal disorders) | 0 | 1
Periodontitis (Gastrointestinal disorders) | 0 | 1
Asthenia (General disorders) | 27 | 23
Chills (General disorders) | 1 | 0
Discomfort (General disorders) | 1 | 0
Disease progression (General disorders) | 50 | 43
Extravasation (General disorders) | 1 | 0
Fatigue (General disorders) | 23 | 29
Gait disturbance (General disorders) | 1 | 1
General physical health deterioration (General disorders) | 3 | 7
Infusion site erythema (General disorders) | 1 | 0
Injection site reaction (General disorders) | 1 | 0
Malaise (General disorders) | 2 | 0
Mucosal inflammation (General disorders) | 4 | 5
Oedema (General disorders) | 3 | 0
Oedema peripheral (General disorders) | 5 | 1
Pain (General disorders) | 2 | 6
Pyrexia (General disorders) | 5 | 3
Thirst (General disorders) | 1 | 0
Ulcer (General disorders) | 1 | 0
Catheter site pain (General disorders) | 0 | 1
Chest pain (General disorders) | 0 | 3
Influenza like illness (General disorders) | 0 | 1
Infusion related reaction (General disorders) | 0 | 2
Non-cardiac chest pain (General disorders) | 0 | 2
Performance status decreased (General disorders) | 0 | 1
Suprapubic pain (General disorders) | 0 | 2
Hepatic failure (Hepatobiliary disorders) | 1 | 0
Hepatic pain (Hepatobiliary disorders) | 1 | 1
Hepatotoxicity (Hepatobiliary disorders) | 2 | 0
Jaundice (Hepatobiliary disorders) | 4 | 0
Jaundice cholestatic (Hepatobiliary disorders) | 2 | 0
Bile duct obstruction (Hepatobiliary disorders) | 0 | 2
Cholecystitis (Hepatobiliary disorders) | 0 | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 2 | 3
Seasonal allergy (Immune system disorders) | 1 | 0
Drug hypersensitivity (Immune system disorders) | 0 | 1
Gastroenteritis viral (Infections and infestations) | 1 | 0
Gingival abscess (Infections and infestations) | 1 | 0
Infection (Infections and infestations) | 1 | 3
Klebsiella bacteraemia (Infections and infestations) | 1 | 0
Lower respiratory tract infection (Infections and infestations) | 2 | 0
Nasopharyngitis (Infections and infestations) | 3 | 0
Onychomycosis (Infections and infestations) | 1 | 0
Paronychia (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 1 | 1
Pyelonephritis (Infections and infestations) | 1 | 0
Sinusitis (Infections and infestations) | 1 | 1
Tooth abscess (Infections and infestations) | 2 | 0
Upper respiratory tract infection (Infections and infestations) | 2 | 2
Urinary tract infection (Infections and infestations) | 11 | 7
Abdominal sepsis (Infections and infestations) | 0 | 1
Bacteraemia (Infections and infestations) | 0 | 1
Bronchitis (Infections and infestations) | 0 | 1
Escherichia infection (Infections and infestations) | 0 | 1
Localised infection (Infections and infestations) | 0 | 1
Respiratory tract infection (Infections and infestations) | 0 | 1
Bone fissure (Injury, poisoning and procedural complications) | 1 | 0
Contrast media reaction (Injury, poisoning and procedural complications) | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 1 | 0
Excoriation (Injury, poisoning and procedural complications) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 2 | 0
Hand fracture (Injury, poisoning and procedural complications) | 1 | 0
Joint injury (Injury, poisoning and procedural complications) | 1 | 0
Procedural pain (Injury, poisoning and procedural complications) | 1 | 0
Skeletal injury (Injury, poisoning and procedural complications) | 2 | 0
Spinal cord injury cauda equina (Injury, poisoning and procedural complications) | 1 | 0
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 1 | 0
Anastomotic leak (Injury, poisoning and procedural complications) | 0 | 1
Fracture (Injury, poisoning and procedural complications) | 0 | 1
Alanine aminotransferase increased (Investigations) | 3 | 4
Aspartate aminotransferase increased (Investigations) | 3 | 4
Blood albumin decreased (Investigations) | 1 | 0
Blood alkaline phosphatase increased (Investigations) | 5 | 5
Blood bilirubin increased (Investigations) | 2 | 3
Blood creatine increased (Investigations) | 1 | 0
Blood creatine phosphokinase increased (Investigations) | 1 | 0
Blood creatinine increased (Investigations) | 5 | 5
Blood lactate dehydrogenase increased (Investigations) | 1 | 0
Gamma-glutamyltransferase increased (Investigations) | 9 | 11
Platelet count decreased (Investigations) | 1 | 1
Transaminases increased (Investigations) | 2 | 0
Weight decreased (Investigations) | 10 | 17
White blood cell count decreased (Investigations) | 1 | 0
Amino acid level increased (Investigations) | 0 | 1
Breath sounds abnormal (Investigations) | 0 | 1
Glomerular filtration rate decreased (Investigations) | 0 | 1
International normalised ratio increased (Investigations) | 0 | 2
Alkalosis (Metabolism and nutrition disorders) | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 34 | 37
Dehydration (Metabolism and nutrition disorders) | 4 | 9
Diabetes mellitus (Metabolism and nutrition disorders) | 2 | 0
Hypercholesterolaemia (Metabolism and nutrition disorders) | 1 | 0
Hypercreatininaemia (Metabolism and nutrition disorders) | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 22 | 27
Hyperuricaemia (Metabolism and nutrition disorders) | 1 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 2 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 2
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 2
Gout (Metabolism and nutrition disorders) | 0 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 | 3
Back pain (Musculoskeletal and connective tissue disorders) | 16 | 12
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Coccydynia (Musculoskeletal and connective tissue disorders) | 1 | 1
Groin pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Limb discomfort (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscle haemorrhage (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 5 | 7
Muscular weakness (Musculoskeletal and connective tissue disorders) | 2 | 2
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 2 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 7 | 3
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 2
Osteoporotic fracture (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 7 | 1
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Tendonitis (Musculoskeletal and connective tissue disorders) | 1 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 2
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 3
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 | 2
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Ageusia (Nervous system disorders) | 1 | 0
Aphonia (Nervous system disorders) | 1 | 0
Cerebral haemorrhage (Nervous system disorders) | 1 | 0
Cognitive disorder (Nervous system disorders) | 1 | 1
Dizziness (Nervous system disorders) | 3 | 3
Dysgeusia (Nervous system disorders) | 2 | 3
Headache (Nervous system disorders) | 6 | 8
Hypoaesthesia (Nervous system disorders) | 1 | 0
Intention tremor (Nervous system disorders) | 1 | 0
Lethargy (Nervous system disorders) | 12 | 6
Peripheral sensory neuropathy (Nervous system disorders) | 1 | 0
Presyncope (Nervous system disorders) | 1 | 0
Sinus headache (Nervous system disorders) | 1 | 0
Hepatic encephalopathy (Nervous system disorders) | 0 | 1
Neurotoxicity (Nervous system disorders) | 0 | 1
Peripheral motor neuropathy (Nervous system disorders) | 0 | 1
Transient ischaemic attack (Nervous system disorders) | 0 | 1
Tremor (Nervous system disorders) | 0 | 1
Anxiety (Psychiatric disorders) | 1 | 1
Confusional state (Psychiatric disorders) | 3 | 7
Depressed mood (Psychiatric disorders) | 1 | 0
Depression (Psychiatric disorders) | 2 | 4
Food aversion (Psychiatric disorders) | 1 | 0
Insomnia (Psychiatric disorders) | 5 | 4
Bladder dilatation (Renal and urinary disorders) | 1 | 0
Choluria (Renal and urinary disorders) | 2 | 0
Dysuria (Renal and urinary disorders) | 2 | 2
Haematuria (Renal and urinary disorders) | 5 | 3
Hydronephrosis (Renal and urinary disorders) | 1 | 1
Nephropathy toxic (Renal and urinary disorders) | 1 | 0
Nocturia (Renal and urinary disorders) | 1 | 0
Pollakiuria (Renal and urinary disorders) | 1 | 3
Polyuria (Renal and urinary disorders) | 1 | 0
Renal disorder (Renal and urinary disorders) | 1 | 0
Renal failure (Renal and urinary disorders) | 3 | 1
Renal failure acute (Renal and urinary disorders) | 4 | 2
Bladder spasm (Renal and urinary disorders) | 0 | 1
Glycosuria (Renal and urinary disorders) | 0 | 1
Proteinuria (Renal and urinary disorders) | 0 | 3
Urinary incontinence (Renal and urinary disorders) | 0 | 1
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 | 0
Ejaculation disorder (Reproductive system and breast disorders) | 1 | 0
Erectile dysfunction (Reproductive system and breast disorders) | 1 | 0
Oedema genital (Reproductive system and breast disorders) | 1 | 0
Pelvic pain (Reproductive system and breast disorders) | 2 | 4
Vaginal discharge (Reproductive system and breast disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 7 | 7
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 3 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 8 | 6
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3 | 2
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 3
Increased viscosity of bronchial secretion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 3
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 3
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Painful respiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Alopecia (Skin and subcutaneous tissue disorders) | 2 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 2 | 2
Erythema (Skin and subcutaneous tissue disorders) | 2 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 1
Macule (Skin and subcutaneous tissue disorders) | 1 | 0
Nail toxicity (Skin and subcutaneous tissue disorders) | 1 | 0
Onychoclasis (Skin and subcutaneous tissue disorders) | 1 | 1
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 2 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 9 | 5
Rash (Skin and subcutaneous tissue disorders) | 4 | 6
Rash macular (Skin and subcutaneous tissue disorders) | 1 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 0
Drug eruption (Skin and subcutaneous tissue disorders) | 0 | 1
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 | 1
Hypoaesthesia facial (Skin and subcutaneous tissue disorders) | 0 | 1
Psoriasis (Skin and subcutaneous tissue disorders) | 0 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 1
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 1
Deep vein thrombosis (Vascular disorders) | 1 | 0
Hypertension (Vascular disorders) | 2 | 6
Flushing (Vascular disorders) | 0 | 2
Hypotension (Vascular disorders) | 0 | 1
Intra-abdominal haematoma (Vascular disorders) | 0 | 1
Superior vena caval occlusion (Vascular disorders) | 0 | 1
Eye disorder (Eye disorders) | 1 | 0
Eye pain (Eye disorders) | 1 | 1
Periorbital oedema (Eye disorders) | 1 | 0
Ocular hyperaemia (Eye disorders) | 0 | 2
Vision blurred (Eye disorders) | 0 | 1
Cushingoid (Endocrine disorders) | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.